CLINICAL TRIAL: NCT03264092
Title: Comparison of Three Different Tissue Acquisition Techniques During Endoscopic Ultrasound-guide Fine Needle Biopsies of Solid Tumors: A Randomized Single Blind Clinical Trial.
Brief Title: Comparison of Three Tissue Acquiring Techniques During EUS Guided Biopsies of Solid Tumors.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary analysis of the results showed no statistically significant difference
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Antonio Mendoza-Ladd, Assistant Professor of Medicine, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E17118
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wet suction (Experimental): This arm will include all the patients that will get an endoscopic ultrasound guided fine needle biopsy done with the wet suction technique
  Interventions: Procedure: Endoscopic ultrasound guided fine needle biopsy
- Dry suction (Experimental): This arm will include all the patients that will get and endoscopic ultrasound guided fine needle biopsy done with the dry suction technique
  Interventions: Procedure: Endoscopic ultrasound guided fine needle biopsy
- Slow pull (Experimental): This arm will include all the patients that will get an endoscopic ultrasound guided fine needle biopsy done with the slow pull technique
  Interventions: Procedure: Endoscopic ultrasound guided fine needle biopsy

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided fine needle biopsy — Using the echoendoscope the lesion is identified and the needle is inserted in it to obtain a biopsy also under sonographic guidance

SUMMARY:
The study's aim is to prospectively compare three different tissue acquisition techniques during EUS guided solid lesions biopsies.

DETAILED DESCRIPTION:
Endoscopic ultrasound guided fine-needle aspiration (EUS-FNA) has been used since 1990's for the diagnosis and staging of esophageal, gastric, duodenal, pancreatobiliary, rectal mediastinal lesions and intra-abdominal lymphadenopathy. Studies have shown a variable range of specimen adequacy when performing pancreatic biopsies with the standard fine needle aspiration (FNA) needles with this modality. There are several factors that affect the overall diagnostic yield of this procedure, such as endosonographer experience, presence of cytopathologist during the procedure, the needle diameter and the number of passes. In this study we will compare the yield of recently available fine biopsy needles (FNB) using three different techniques to obtain samples from solid lesions. The three techniques to be compared in this study are: stylet slow pull (SP) vs dry suction (DS) vs wet suction (WS).

wall cells.

In the "suction technique" the stylet of the needle can be left in place or removed before puncturing the lesion. Once the needle is inside the target, negative pressure is applied through a 10 or 20 cc syringe connected to the needle.

The wet suction technique consists of flushing of the needle with 5 ml of saline solution to replace the column of air within the lumen of needle with saline solution before needle aspiration. Once the needle is flushed, negative pressure is applied with a 10 or 20 cc syringe connected to the needle.

In the slow pull technique, the stylet is left in place in the needle and is slightly retracted prior to puncturing the lesion. Once the needle is inside the target, the stylet is pushed completely into the needle to remove any contaminant cells and several back and forth movements are done while slowly withdrawing the stylet.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18-80 years old
2. Sex: male or female
3. Patients who require EUS and tissue sampling of solid solid lesions (size >1 cm) anywhere in the following locations: lymph nodes, stomach, esophagus, colon, small intestine, pancreas, liver, spleen or kidney.
4. Patients who are able to give consent

Exclusion Criteria:

1. Pregnant female
2. Coagulation disorders (platelets < 50,000/mm3, INR > 2)
3. Patients with acute pancreatitis in the immediate 2 weeks prior to the procedure.
4. Cardiorespiratory dysfunction that precludes sedation.
5. Unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Mendoza Ladd, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech university Health Sciences Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamao K, Sawaki A, Mizuno N, Shimizu Y, Yatabe Y, Koshikawa T. Endoscopic ultrasound-guided fine-needle aspiration biopsy (EUS-FNAB): past, present, and future. J Gastroenterol. 2005 Nov;40(11):1013-23. doi: 10.1007/s00535-005-1717-6. PMID 16322944
- [Background] Puri R, Vilmann P, Saftoiu A, Skov BG, Linnemann D, Hassan H, Garcia ES, Gorunescu F. Randomized controlled trial of endoscopic ultrasound-guided fine-needle sampling with or without suction for better cytological diagnosis. Scand J Gastroenterol. 2009;44(4):499-504. doi: 10.1080/00365520802647392. PMID 19117242
- [Derived] Mendoza Ladd A, Casner N, Cherukuri SV, Garcia C, Padilla O, Dwivedi A, Hakim N. Fine Needle Biopsies of Solid Pancreatic Lesions: Tissue Acquisition Technique and Needle Design Do Not Impact Specimen Adequacy. Dig Dis Sci. 2022 Sep;67(9):4549-4556. doi: 10.1007/s10620-021-07316-4. Epub 2021 Dec 2. PMID 34859313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early given the difficulty we experienced enrolling patients.
Groups:
- Wet Suction: This arm included all the patients that got an endoscopic ultrasound guided fine needle biopsy done with the wet suction technique=17
  Endoscopic ultrasound guided fine needle biopsy: Using the echoendoscope the lesion is identified and the needle is inserted in it to obtain a biopsy also under sonographic guidance
- Dry Suction: This arm included all the patients that got and endoscopic ultrasound guided fine needle biopsy done with the dry suction technique=20
  Endoscopic ultrasound guided fine needle biopsy: Using the echoendoscope the lesion is identified and the needle is inserted in it to obtain a biopsy also under sonographic guidance
- Slow Pull: This arm included all the patients that got an endoscopic ultrasound guided fine needle biopsy done with the slow pull technique=17
  Endoscopic ultrasound guided fine needle biopsy: Using the echoendoscope the lesion is identified and the needle is inserted in it to obtain a biopsy also under sonographic guidance
Period: Overall Study
Arm/Group | Wet Suction | Dry Suction | Slow Pull
Started | 17 | 20 | 18
Completed | 17 | 20 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wet Suction | Dry Suction | Slow Pull | Total
Number analyzed (Participants) | 17 | 20 | 18 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (13) | 64 (14) | 66 (10) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 6 | 23
  Male | 7 | 13 | 12 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 17 | 15 | 45
  Not Hispanic or Latino | 4 | 3 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 18 | 55

OUTCOME MEASURES:

1. Primary Outcome: Cellularity of Specimens Obtained by Each Individual Technique Based on Cellularity Score
Description: 0: inadequate
  1. limited cytological dx
  2. adquate cytological dx
  3. limited histological dx
  4. adequate histological dx with low quality
  5. adequate histological dx with high quality
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Wet Suction: This arm describes the mean cellularity score obtained with the wet suction technique.
- Dry Suction: This arm describes the mean cellularity score obtained with the dry suction technique.
- Slow Pull: This arm describes the mean cellularity score obtained with the slow pull technique.
Arm/Group | Wet Suction | Dry Suction | Slow Pull
Number analyzed (Participants) | 17 | 20 | 18
units on a scale | 2.94 (0.75) | 3.55 (0.76) | 3.28 (0.89)
Statistical Analysis 1: Comparison: Wet Suction vs Dry Suction vs Slow Pull; Test type: Other — This was just a comparative study. No superiority, equivalence or non inferiority analysis was performed; p = 0.18, Fisher Exact

2. Secondary Outcome: Blood Contamination Score of Each Specimen Obtained
Description: This is based on the following scale
  1. Blood present
  2. Blood clots present
Time Frame: 2 hours
Measure: Number; unit: participants
Groups:
- Wet Suction: This arm describes the number of subjects with each specific blood contamination score from all of those obtained with the wet suction technique.
- Dry Suction: This arm describes the number of subjects with each specific blood contamination score from all of those obtained with the dry suction technique.
- Slow Pull: This arm describes the number of subjects with each specific blood contamination score from all of those obtained with the slow pull technique.
Arm/Group | Wet Suction | Dry Suction | Slow Pull
Number analyzed (Participants) | 17 | 20 | 18
participants
  Blood present | 17 | 19 | 18
  Blood clot present | 0 | 1 | 0
Statistical Analysis 1: Comparison: Wet Suction vs Dry Suction vs Slow Pull; Test type: Other — This was just a comparative study. No superiority, equivalence or non inferiority analysis was performed; p = 0.41, Fisher Exact

3. Secondary Outcome: Number of Participants Stratified Per the Number of Diagnostic Passes Required
Description: This indicates which out of the 3 passes provided enough tissue for diagnosis. If after 3 passes not enough tissue was obtained, the doctor was free to use the technique of his preference outside of the protocol.
Time Frame: 2 hours
Population: Diagnostic passes 4 and above were considered outside of protocol
Measure: Number; unit: participants
Groups:
- Wet Suction: This arm included all the patients that got an endoscopic ultrasound guided fine needle biopsy done with the wet suction technique=17 subjects
- Dry Suction: This arm included all the patients that got an endoscopic ultrasound guided fine needle biopsy done with the dry suction technique=20 subjects
- Slow Pull: This arm included all the patients that got an endoscopic ultrasound guided fine needle biopsy done with the slow pull technique=18 subjects
Arm/Group | Wet Suction | Dry Suction | Slow Pull
Number analyzed (Participants) | 17 | 20 | 18
participants
  Diagnostic pass 1 | 6 | 11 | 7
  Diagnostic pass 2 | 7 | 5 | 4
  Diagnostic pass 3 | 3 | 3 | 6
  Diagnostic pass 4 | 1 | 0 | 0
  Diagnostic pass 5 | 0 | 1 | 0
  Diagnostic pass 6 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Wet Suction vs Dry Suction vs Slow Pull; Test type: Other — This was just a comparative study. No superiority, equivalence or non inferiority analysis was performed; p = 0.45, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 hours
Description: Adverse events evaluated in this study were: bleeding, bowel perforation and hemodynamic instability. The definitions of these adverse events are similar to the ones established by clinicaltrials.gov
Groups:
- Dry Suction: This arm included all the patients that got and endoscopic ultrasound guided fine needle biopsy done with the dry suction technique=20 subjects
- Slow Pull: This arm included all the patients that got an endoscopic ultrasound guided fine needle biopsy done with the slow pull technique=18 subjects
  \
Arm/Group | Wet Suction | Dry Suction | Slow Pull
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 3/20 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wet Suction (N=17) | Dry Suction (N=20) | Slow Pull (N=18)
Bleeding (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) — Bleeding from the puncture site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03264092/Prot_SAP_000.pdf